CLINICAL TRIAL: NCT00728533
Title: The Rationale of the Study is to Demonstrate That Degarelix Given at Three-month Dosing Intervals Will Produce and Maintain Androgen Deprivation in Prostate Cancer Patients Through Immediate and Prolonged Testosterone Suppression, and to Provide Confirmatory Evidence of the Safety of Degarelix.
Brief Title: Open-Label, Randomised Parallel-Group Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to awaiting data from Phase II study.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS26; 2007-006055-39
Record Dates: First submitted 2008-01-18; First posted 2008-08-06 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer requiring Androgen Ablation Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): * Starting dose of 240 mg (40 mg/mL) will be given on Day 0.
  * Maintenance doses of 360 mg (60 mg/mL) will be given after 1, 4, 7, and 10 months
  Interventions: Drug: Degarelix
- 2 (Experimental): * Starting dose of 240 mg (40 mg/mL) will be given on Day 0.
  * Maintenance doses of 480 mg (60 mg/mL) will be given after 1, 4, 7, and 10 months.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Prostate Cancer - Degarelix powder and solvent for suspension for injection. Three-month depot in two dosing regimens.
  Arms: 1
Drug: Degarelix — Prostate Cancer - Degarelix powder and solvent for suspension for injection. Three-month depot in two dosing regimens.
  Arms: 2

SUMMARY:
An Open-Label, Multi-Centre, Randomised Parallel-Group Study, Investigating Efficacy and Safety of Different Degarelix Three-Month Dosing Regimens in Patients with Prostate Cancer Requiring Androgen Ablation Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged 18 years or older, with a histologically proven prostate cancer of all stages in whom endocrine treatment is indicated.
* Screening testosterone level above the lower limit of normal range, globally defined as > 2.2 ng/mL.
* Screening PSA level of =2 ng/mL. ECOG score of =2.
* Life expectancy of at least one year.

CRITERIA FOR EVALUATION:

Primary endpoint:

* Probability of testosterone at castrate level (=0.5 ng/mL) from Day 28 through Day 364.

Secondary endpoints:

* Probability of testosterone at castrate level (=0.5 ng/mL) from Day 56 through Day 364.
* Serum levels of testosterone, LH, FSH, and PSA over time.
* Time to PSA failure - defined as two consecutive increases of 50%, and at least 5 ng/mL, compared to nadir.
* Plasma levels of degarelix over time.
* Frequency and severity of adverse events.
* Clinically significant changes in laboratory safety parameters.
* Clinically significant changes in physical examinations, ECGs, vital signs, and body weight.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To demonstrate efficacy of degarelix in achieving and maintaining testosterone suppression at castrate levels (=0.5 ng/mL) during one year of treatment in prostate cancer patients. | 3-month

SECONDARY OUTCOMES:
To evaluate testosterone, PSA, LH, and FSH responses during one year of treatment. | 3-month
To evaluate pharmacokinetic response. | 3-month
To compare safety and tolerability profiles of different degarelix three-month dosing regimens. | 3-month

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals